CLINICAL TRIAL: NCT01007734
Title: Factors Determining Quality of Life Related to Respiratory Status According to Gender of COPD Patients Followed by a Pneumologist
Brief Title: Factors Determining Quality of Life Related to Respiratory Status According to Gender of Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: VITALITE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Castaigne, Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-RFR-DUM-2009/1
Record Dates: First submitted 2009-10-31; First posted 2009-11-04 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Quality of life; COPD patients; Evaluation According to Gender the Determining Independent Factors of Quality of Life Related to Respiratory Status of Patient With Moderate to Severe COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this study is to evaluate with sufficient precision and according to gender the determining independent factors of quality of life related to respiratory status of patient with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient who has a clinical visit for their usual follow-up.
* patient with COPD with at least a three month follow up

Exclusion Criteria:

* Current or history of asthma
* Current participation in an interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First 3 consecutive adults with COPD with at least a three month follow up, seen by pneumologist
Sampling Method: Probability Sample
Enrollment: 449 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To evaluate with sufficient precision and according to gender the determining independent factors of quality of life related to respiratory status of patient with moderate to severe COPD

CONTACTS AND LOCATIONS:
Overall Officials: Alain Alain Castaigne, Medical Director, Study Director — AstraZeneca
Locations (178):
- France (178):
  - Research Site, Abbeville
  - Research Site, Agde
  - Research Site, Agen
  - Research Site, Aix-en-Provence
  - Research Site, Ajaccio
  - Research Site, Albi
  - Research Site, Alençon
  - Research Site, Alès
  - Research Site, Ambilly
  - Research Site, Amelie Les Bains Palalda
  - Research Site, Amiens
  - Research Site, Angers
  - Research Site, Angoulême
  - Research Site, Annecy
  - Research Site, Antibes
  - Research Site, Antony
  - Research Site, Armentières
  - Research Site, Auch
  - Research Site, Bagneux
  - Research Site, Bastia
  - Research Site, Bayonne
  - Research Site, Beauvais
  - Research Site, Belfort
  - Research Site, Berck
  - Research Site, Besançon
  - Research Site, Beuvry
  - Research Site, Béthune
  - Research Site, Béziers
  - Research Site, Bois-Guillaume
  - Research Site, Bonneville
  - Research Site, Bordeaux
  - Research Site, Bourges
  - Research Site, Bourgoin
  - Research Site, Brest
  - Research Site, Briey
  - Research Site, Brive-la-Gaillarde
  - Research Site, Cachan
  - Research Site, Caen
  - Research Site, Cagnes-sur-Mer
  - Research Site, Calais
  - Research Site, Cambo-les-Bains
  - Research Site, Cambrai
  - Research Site, Cannes
  - Research Site, Castelnau-le-Lez
  - Research Site, Cavaillon
  - Research Site, Challans
  - Research Site, Chalon-sur-Saône
  - Research Site, Chamalières
  - Research Site, Chambéry
  - Research Site, Charleville-Mézières
  - Research Site, Châlons-en-Champagne
  - Research Site, Cherbourg Octeville
  - Research Site, Cholet
  - Research Site, Clermont-Ferrand
  - Research Site, Cluses
  - Research Site, Cognac
  - Research Site, Colmar
  - Research Site, Corbeil-Essonnes
  - Research Site, Courbevoie
  - Research Site, Croix
  - Research Site, Denain
  - Research Site, Divion
  - Research Site, Écully
  - Research Site, Épernay
  - Research Site, Facture
  - Research Site, Figeac
  - Research Site, Fleury-les-Aubrais
  - Research Site, Foix
  - Research Site, Fontenay-le-Comte
  - Research Site, Fréjus
  - Research Site, Gap
  - Research Site, Givors
  - Research Site, Grande-Synthe
  - Research Site, Grenoble
  - Research Site, Guingamp
  - Research Site, Hagondange
  - Research Site, Herblay-sur-Seine
  - Research Site, Hyères
  - Research Site, Istres
  - Research Site, Jonzac
  - Research Site, Juan-les-Pins
  - Research Site, Juvisy-sur-Orge
  - Research Site, La Ferté-Bernard
  - Research Site, La Rochelle
  - Research Site, La Teste-de-Buch
  - Research Site, Lagny-sur-Marne
  - Research Site, Laon
  - Research Site, Le Cannet
  - Research Site, Le Chesnay
  - Research Site, Lens
  - Research Site, Lège-Cap-Ferret
  - Research Site, Libourne
  - Research Site, Liévin
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, LIsle-dEspagnac
  - Research Site, Lodève
  - Research Site, Lorient
  - Research Site, Lormont
  - Research Site, Lutterbach
  - Research Site, Lyon
  - Research Site, Maisons-Alfort
  - Research Site, Maisons-Laffitte
  - Research Site, Mandelieu-la-Napoule
  - Research Site, Marignane
  - Research Site, Marly-le-Roi
  - Research Site, Marmande
  - Research Site, Marseille
  - Research Site, Melun
  - Research Site, Mende
  - Research Site, Millau
  - Research Site, Molsheim
  - Research Site, Montauban
  - Research Site, Montbéliard
  - Research Site, Montfermeil
  - Research Site, Montgeron
  - Research Site, Montigny-lès-Metz
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Nans-les-Pins
  - Research Site, Nantes
  - Research Site, Narbonne
  - Research Site, Nevers
  - Research Site, Nice
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Nogent-sur-Marne
  - Research Site, Ollioules
  - Research Site, Oloron-Sainte-Marie
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Perpignan
  - Research Site, Pessac
  - Research Site, Pézenas
  - Research Site, Poitiers
  - Research Site, Pontault-Combault
  - Research Site, Pontivy
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Royan
  - Research Site, Rueil-Malmaison
  - Research Site, Saint-André-les-Vergers
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Denis
  - Research Site, Saint-Estève
  - Research Site, Saint-Etienne
  - Research Site, Saint-Girons
  - Research Site, Saint-Jean-de-Maurienne
  - Research Site, Saint-Julien-de-Raz
  - Research Site, Saint-Martin-Boulogne
  - Research Site, Saint-Martin-d'Hères
  - Research Site, Saint-Orens-de-Gameville
  - Research Site, Saint-Quentin
  - Research Site, Sarlat-la-Canéda
  - Research Site, Sens
  - Research Site, Sélestat
  - Research Site, St-Malo
  - Research Site, St.-Jean
  - Research Site, Ste Clotilde Cedex
  - Research Site, Strasbourg
  - Research Site, Taden
  - Research Site, Tergnier
  - Research Site, Thionville
  - Research Site, Thonon-les-Bains
  - Research Site, Thouars
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Tours
  - Research Site, Valence
  - Research Site, Valenciennes
  - Research Site, Vénissieux
  - Research Site, Vienne
  - Research Site, Vierzon
  - Research Site, Villefranche-de-Lauragais
  - Research Site, Villefranche-sur-Saône
  - Research Site, Villeurbanne